CLINICAL TRIAL: NCT01795001
Title: The Molecular Pathogenesis of Late-onset Fuchs' Endothelial Corneal Dystrophy
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); Funds for Research in Ophthalmology, Belgium (Unknown); Mieke Perdaens fund for Eye Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: S55133
Record Dates: First submitted 2013-01-30; First posted 2013-02-20 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Fuchs' Endothelial Dystrophy
Keywords: pathophysiology
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Non-interventional study on corneal endothelium, anterior eye chamber fluid and paraffin-embedded corneal tissue, using molecular techniques to identify and characterise the molecular players involved in the pathogenesis of FECD.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- late-onset FECD: tissue samples from patients with late-onset Fuchs' endothelial corneal dystrophy (FECD)
  Interventions: Other: No intervention
- normal control: tissue samples from patients with normal corneas
  Interventions: Other: No intervention
- non-FECD edematous control: tissue samples from patients with corneal edema but without FECD
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The purpose of this study is to gain further insights into the molecular pathogenesis of Fuchs' endothelial corneal dystrophy (FECD), to identify targets for potential specific drug therapy.

ELIGIBILITY:
Inclusion Criteria:

* FECD
* normal corneas (including enucleations for uveal melanoma)
* non-FECD oedematous corneas

Exclusion Criteria:

* prior irradiation therapy for uveal melanoma
* corneal extension of uveal melanoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Fuchs' Endothelial Corneal Dystrophy (FECD), normal control patients, and patients with non-Fuchs edematous corneas; in university hospital setting.
Sampling Method: Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2012-10; Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
cytokine levels | at time of prelevation (once, no intervention)
  dosage of cytokine levels in aqueous humour (exploratory, non-interventional study)
gene expression levels | at time of prelevation (once, no intervention)
  microarray expression analysis, reverse transcriptase - quantitative polymerase chain reaction (RT-qPCR), RNA-sequencing (exploratory, non-interventional study)
protein content | at time of prelevation (once, no intervention)
  immunohistochemistry and immunofluorescence

CONTACTS AND LOCATIONS:
Overall Officials: Joost J van den Oord, MD, PhD, Principal Investigator — KU Leuven
Locations (1):
- Department of Translational Cell and Tissue Research - campus Sint-Raf - UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
MEA and RT-qPCR data have been deposited in NCBI's Gene Expression Omnibus and are accessible through the Gene Expression Omnibus Series accession number GSE75676.
Supporting Information: Study Protocol
Time Frame: Data already available.
URL: https://www.ncbi.nlm.nih.gov/geo/query/acc.cgi?acc=GSE75676